CLINICAL TRIAL: NCT06077526
Title: Alleviating Burden of Chronic Musculoskeletal Pain in the Emergency Department: P.E.A.K. Rx Feasibility Trial
Brief Title: Alleviating Burden of Chronic Musculoskeletal Pain in the Emergency Department
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bridgewater College (Other)
Responsible Party: Principal Investigator, Michael Ray, Assistant Professor, Bridgewater College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-010
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: musculoskeletal
MeSH Terms: conditions — Chronic Pain | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Upon recruitment and completion of informed consent, participants will be randomly assigned following a stratified randomization schedule to either Group A or B using online randomization software. A stratified randomization schedule was selected to balance the group assignments based on the covariate of sex. A team member who will have no contact with participants will obtain and employ the randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - P.E.A.K. Rx (Experimental): Group A intervention, P.E.A.K. Rx, will be supervised and directed by healthcare clinicians, known as Pain Coaches. P.E.A.K. Rx will involve 2 meetings per week of pain education + physical activity.
  Interventions: Behavioral: P.E.A.K. Rx
- Control - Usual Care (Active Comparator): Group B will receive the community hospital's usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: P.E.A.K. Rx — Pain Education + Physical Activity Group Based Intervention
  Other Names: Rehabilitation Therapy
  Arms: Experimental - P.E.A.K. Rx
Other: Usual Care — Participants will receive the community hospital's usual care.
  Arms: Control - Usual Care

SUMMARY:
Chronic musculoskeletal pain (CMP) and lack of physical activity often co-exist, contributing to increased disability, non-communicable diseases (e.g., obesity, diabetes, hypertension), psychological comorbidity (e.g., anxiety and depression), and healthcare utilization and costs [1-6]. Many individuals with CMP seek assistance at emergency departments (ED). ED overuse has been an ongoing concern, with 1-in-5 Americans presenting to the ED at least once each year [7]. Of these visits, 24 million are for adults seeking help for chronic pain, with an additional 12 million due to exacerbations of an existing chronic pain condition [8]. In 2021, the fourth most common reason for seeking care in the ED related to a primary diagnosis involving the musculoskeletal system, with an estimated 9.5 million visits [9]. Most ED visits result in a 'treat and release' approach, potentially disrupting continuity of care and resulting in follow-up ED visits [10]. These ED visits for chronic pain are indicative of accessibility problems to community-based primary and preventative care, compounded by limited or no health insurance coverage [10]. Based on the Emergency Medical Treatment and Labor Act, EDs are required to stabilize all patients regardless of ability to pay [10]. To alleviate the burden of CMP on patients and EDs, improve access to quality healthcare, and mitigate initial and repeat ED visits, alternative options are required. Here we propose a novel group-based intervention involving pain education (PE) and physical activity (PA) implemented in CMP patients presenting to the ED of a community level hospital. The investigators will recruit 60 adults from a community hospital located in the Shenandoah Valley region of Virginia; participants will be randomized to either Pain Education and Active Knowledge (P.E.A.K.) Rx (24 sessions of group PE+ + PA) or usual care. Research assessments are conducted with both groups at study entry (baseline), 8-weeks, 3-months, and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Sedentary (e.g., not meeting PA guidelines, assessed by ACSM PA vitals)
* English speaking and reading comprehension
* Not currently pregnant
* Diagnosed with CMP based on electronic health record:

  * Non-red flag presentation (e.g., red flags: current fracture, malignancy, infection, vascular issues, or in need of surgical intervention).
  * Persistent or recurrent pain for 3+ months, with at least moderate pain intensity level (Visual Analog Scale of 40/100)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Quantitative metric of an individual's pain on a numerical scale. Scores range from 0 - 100, where 0 means no pain and 100 means maximum pain.
  1-30 = mild 31-69 = moderate 70-100 = severe MCID of 12 point change [60].

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Quantitative metric asking 17 questions using a 4-point Likert scale regarding a participant's fear and avoidance of movement. Scores range from 17 to 68, where 17 means no kinesiophobia and higher scores indicate increasing severity of kinesiophobia. Scores ≥ 37 indicate kinesiophobia. MCID of 7.5-9 points [61].
Pain Catastrophizing Scale | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  13-item quantitative metric assessing participant's catastrophic thinking about their pain experience, contributing to rumination, magnification, and learned helplessness. Utilizes 4-item scale to assess frequency of particular thoughts, 0 = not at all to 4 = all the time. Total score ranges from 0 - 52. Score ≥ 30 indicates catastrophizing.
  MCID of 11 points for those considered to be engaging in catastrophic thinking (baseline score >30 points) [62].
Patient Specific Functional Scale (PSFS) | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Assesses impact of pain on participant's function by identification of difficult or unable to perform activities. 11-point Likert scale ranks participant's current level of difficulty for each activity (0 = unable to perform, 10 = able to perform activity at same level before injury or problem).
  Assess improvement in function of valued activities post intervention. MCID is categorized:
  Small change = 1.3 Medium change = 2.3 Large change = 2.7 [63].
Saltin-Grimby physical activity scale for leisure time physical activity | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Assesses participants perception of their leisure time activities. Describe your exercise and physical exertion in leisure time. If your activity varies much, for example between summer and winter, then give an average. The question refers only to the last year.
  Four different levels:
  "Reading, watching TV, or other sedentary activity," "Walking, cycling, or other forms of exercise at least 4 hours a week (here including walking or cycling to place of work, Sunday walking, etc.)," "Participation in recreational sports, heavy gardening, etc. (note: duration of activity at least 4 hours a week)" and "Participation in hard training or sports competitions, regularly several times a week." 4 levels renamed: "inactive," "low," "moderate," and "vigorous," respectively [65]
36-Item Short Form Health Survey (SF-36) | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  A health-related quality of life survey assessing eight dimensions: physical function, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Scores for each dimension range from 0 (worst level of functioning) to 100 (best level of functioning). Total sore MCID of 4.6 points [64].
Self-report physical exercise | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Exercise assessment through 3 questions on frequency, duration, and intensity, where the respondents will be asked to estimate their weekly average. Frequency question: "How often do you exercise (i.e., walking, skiing, swimming or training/sports)?" Duration question: "For how long (time) do you exercise?" Intensity question "If you exercise-how hard do you exercise?"
  Frequency categories:
  "never", "less than once a week", "once a week", "2 to 3 times a week", or "approximately every day".
  Duration categories:
  "less than 15 minutes", "15 to 29 minutes", "30 to 60 minutes", or "more than 1 hour."
  Intensity categories:
  "Easy-you do not become short-winded or sweaty", "You become short-winded and sweaty", and "Hard-you become exhausted". Categorized as "low", "moderate", and "hard" respectively [65].
Self-report occupational activity | Baseline, post-intervention 8-weeks, 3-months, and 6-months
  Assess occupational physical activity.
  Question: "If you have paid or unpaid work, which statement describes your work best? Response categories:
  "mostly sedentary work (e.g., office work)", "work that requires a lot of walking (e.g., shop assistant, light industrial work)", and "work that requires a lot of walking and lifting (e.g., nursing, construction, or heavy manual labor)".

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ray, DC, MSc, Principal Investigator — Bridgewater College

IPD SHARING:
Plan to Share IPD: Undecided
In line with open science practices, all data and statistical code will be made available following publication of findings (via Open Science Framework).